CLINICAL TRIAL: NCT03161210
Title: Evaluation of Pain Regression in Patients With Myofascial Facial Pain Treated by Dextrose Prolotherapy Versus Local Anesthetic Injections: A Prospective Double-blind Randomized Placebo-controlled Clinical Trial.
Brief Title: Evaluation of Pain Regression in Patients With Myofascial Facial Pain Using Dextrose, Local Anaesthesia and Saline.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Ahmed Mohamed Ammar, Principal Investigator, Internal resident in Oral and Maxillofacial Department, faculty of oral and dental medicine., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28712038800227
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Anesthesia, Local; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dextrose Prolotherapy (Experimental)
  Interventions: Other: Dextrose Prolotherapy
- Local Anaesthetic (Active Comparator)
  Interventions: Other: Local Anaesthesia
- Saline (Placebo Comparator)
  Interventions: Other: Saline

INTERVENTIONS:
Other: Dextrose Prolotherapy — Dextrose is a solution, mixture of dextrose and water.
  Arms: Dextrose Prolotherapy
Other: Local Anaesthesia — A local anaesthetic is a medication that causes reversible absence of pain sensation
  Arms: Local Anaesthetic
Other: Saline — Saline is a control group
  Arms: Saline

SUMMARY:
The aim of this study is to compare the treatment effects of dextrose prolotherapy, saline, and mepivacaine for deactivating myofascial trigger points within the jaw muscles.

ELIGIBILITY:
Inclusion Criteria:

- 1. Presence of active myofacial pains in jaw muscles, previously identified by manual palpation.

2. Age ≥ 18 years. 3. Willingness to follow instructions

Exclusion Criteria:

* 1. Therapeutic intervention for myofascial pain within the past month before the study, such as using of medications for pain control or wearing of occlusal splint.

  2. Clinical conditions such as pregnancy. 3. Medical problems that may interfere with the procedures such as bleeding disorders, trigeminal neuralgia.

  4. Recent facial or neck trauma; medication or adjunctive treatment (eg, physiotherapy) that could not be stopped during the study; or allergy to local anesthetic solutions.

  5. Cognitive impairment or exhibited inadequate cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Patients' subjective pain experience | one year
  Pressure pain threshold (PPT): An algometer will be used to assess PPT. The algometer consists of a 1 cm2 rubber tipped plunger mounted on a force transducer. The pressure will be applied over the examined trigger point. The participants will be instructed to point when the sensation changed from pressure to pain. The mean of three trials will be calculated and used for analysis.

IPD SHARING:
Plan to Share IPD: Undecided